CLINICAL TRIAL: NCT00969319
Title: Effekt-2 - Efficacy and Safety of Long-term Treatment With KOGENATE® FS in Latin America
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 14285; KG0802 (Other: company internal)
Record Dates: First submitted 2009-08-31; First posted 2009-09-01 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Blood Coagulation Disorders; Hemophilia A
Keywords: Octocog alfa; Hemophilia A
MeSH Terms: conditions — Blood Coagulation Disorders; Hemophilia A | interventions — Factor VIII; F8 protein, human; BAY 14-2222

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Biological: Recombinant Factor VIII (Kogenate FS, BAY14-2222)

INTERVENTIONS:
Biological: Recombinant Factor VIII (Kogenate FS, BAY14-2222) — Patients under daily life treatment receiving Kogenate according to local drug information.

SUMMARY:
The aim of this international prospective post-marketing surveillance study is to obtain data on treatment procedures, long-term safety and efficacy and patient acceptance of KOGENATE Bayer/FS in treatment of patients with haemophilia A under daily-life treatment conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of hemophilia A, independent of age, treated with KOGENATE® FS as their only source of FVIII, decision taken by the investigator to administer KOGENATE® FS. For pretreated patients with more than 100 exposure days an inhibitor assessment within three months prior to enrollment should be available; for pretreated patients with less than 100 exposure days an inhibitor assessment at baseline should be available.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of patients with a diagnosis of hemophilia A. Physicians should consult the full prescribing information for KOGENATE® FS before enrolling patients and familiarize themselves with the safety information in the product package label.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2009-09; Primary Completion 2013-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Total consumption of FVIII | After 12 months and after 24 months
Number of bleedings | After 12 months and after 24 months
Kind of bleedings | After 12 months and after 24 months
Continuation of therapy | After 12 months and after 24 months
Overall assessment by the physician | After 12 months and after 24 months

SECONDARY OUTCOMES:
Adverse event collection | After 12 months and after 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- Many Locations, Mexico
- Many Locations, Venezuela